CLINICAL TRIAL: NCT03083093
Title: Identification of CTEPH on Standard Computerised Tomography Pulmonary Angiography Performed in the Work-up of Suspected Pulmonary Embolism
Brief Title: CTEPH Identification an Standard Computerised Tomography Pulmonary Angiography in Pulmonary Embolism Patients
Acronym: InShapeIII
Status: Completed | Type: Observational
Sponsor: Leiden University Medical Center (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Erik Klok, principal investigator, Leiden University Medical Center
Other Study IDs: G17.014
Record Dates: First submitted 2017-03-08; First posted 2017-03-17 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: CTEPH; Pulmonary Embolism; Early Diagnosis
MeSH Terms: conditions — Pulmonary Embolism; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CTEPH patients: the initial CTPA scan will be reviewed in patients diagnosed with CTEPH after an episode of an acute PE
  Interventions: Diagnostic Test: The initial CTPA will be reviewed
- non CTEPH patients: the initial CTPA scan will be reviewed in patients after an episode of an acute PE in whom CTEPH was excluded
  Interventions: Diagnostic Test: The initial CTPA will be reviewed

INTERVENTIONS:
Diagnostic Test: The initial CTPA will be reviewed — The initial CTPA will be reviewed

SUMMARY:
In this study the investigators will evaluate whether more careful reading (than the current standard) of routine computerised tomography pulmonary angiography (CTPA) performed in the clinical work-up of suspected (pulmonary embolism (PE) will differentiate patients with acute PE from those with more chronic or acute on chronic PE, which could be indicative of the presence of chronic thromboembolic pulmonary hypertension (CTEPH)"

DETAILED DESCRIPTION:
The investigators will study 50 consecutive patients diagnosed with CTEPH as well as 50 patients diagnosed with acute PE in whom CTEPH was ruled out 2 years after the PE diagnosis by sequential echocardiography. The cases and controls will be matched based on the right-to-left ventrilcle diameter ratio.

Three experienced thorax radiologists with specific expertise on acute PE and CTEPH will blindly assess the index CTPAs of the study population. In addition to the binominal judgement whether CTEPH signs are already present (or not), the presence of the following items will be scored by all 3 readers independently:

* Webs or bands
* Residual thrombus attached to the vascular wall
* Complete occlusion /retraction
* Mosaic perfusion
* Pulmonary infarct
* Parenchymal bands
* Bronchial arteries
* Right atrial (RA) dilatation
* Right ventricle (RV) dilatation
* Flattening of the septum
* Right ventricle (RV) hypertrophy
* Dilated truncus pulmonalis
* Cardiac signs of pulmonary hypertension (PH)
* Further remarks (free text)

ELIGIBILITY:
Inclusion Criteria:

* patients after an acute PE diagnosed with CTEPH according to current guidelines, patients after an acute PE in whom CTEPH is excluded by follow-up echocardiography
* availability of the CTPA scan of the initial PE episode

Exclusion Criteria:

* CTEPH diagnosis based on other test results than a RHC
* Patients who did not receive anticoagulation after PE diagnosis
* Patients under the age of 18 years old
* Patients in the control group with a follow-up duration of less than 2 years after the index PE episode
* Use of a CTPA scanner with less than 32-detector rows

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The CTPA scans of the following patient populations will be compared. The first group consists of patients with confirmed CTEPH after a prior diagnosis of acute PE. The control group consists of patients with an episode of acute PE in whom CTEPH was excluded after 2 years of follow-up by echocardiography. The CTPA scans of case and control patients will be matched according to the right-to-left ventricule diameter ratio.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: F.A. Klok, MD PhD, Principal Investigator — LUMC department of thormbosis and hemostasis
Locations (1):
- LUMC, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
this has to be planned

REFERENCES:
- [Background] Konstantinides SV. 2014 ESC Guidelines on the diagnosis and management of acute pulmonary embolism. Eur Heart J. 2014 Dec 1;35(45):3145-6. doi: 10.1093/eurheartj/ehu393. No abstract available. PMID 25452462
- [Background] Galie N, Humbert M, Vachiery JL, Gibbs S, Lang I, Torbicki A, Simonneau G, Peacock A, Vonk Noordegraaf A, Beghetti M, Ghofrani A, Gomez Sanchez MA, Hansmann G, Klepetko W, Lancellotti P, Matucci M, McDonagh T, Pierard LA, Trindade PT, Zompatori M, Hoeper M. 2015 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension: The Joint Task Force for the Diagnosis and Treatment of Pulmonary Hypertension of the European Society of Cardiology (ESC) and the European Respiratory Society (ERS): Endorsed by: Association for European Paediatric and Congenital Cardiology (AEPC), International Society for Heart and Lung Transplantation (ISHLT). Eur Respir J. 2015 Oct;46(4):903-75. doi: 10.1183/13993003.01032-2015. Epub 2015 Aug 29. PMID 26318161
- [Background] Pepke-Zaba J, Delcroix M, Lang I, Mayer E, Jansa P, Ambroz D, Treacy C, D'Armini AM, Morsolini M, Snijder R, Bresser P, Torbicki A, Kristensen B, Lewczuk J, Simkova I, Barbera JA, de Perrot M, Hoeper MM, Gaine S, Speich R, Gomez-Sanchez MA, Kovacs G, Hamid AM, Jais X, Simonneau G. Chronic thromboembolic pulmonary hypertension (CTEPH): results from an international prospective registry. Circulation. 2011 Nov 1;124(18):1973-81. doi: 10.1161/CIRCULATIONAHA.110.015008. Epub 2011 Oct 3. PMID 21969018
- [Background] Tunariu N, Gibbs SJ, Win Z, Gin-Sing W, Graham A, Gishen P, Al-Nahhas A. Ventilation-perfusion scintigraphy is more sensitive than multidetector CTPA in detecting chronic thromboembolic pulmonary disease as a treatable cause of pulmonary hypertension. J Nucl Med. 2007 May;48(5):680-4. doi: 10.2967/jnumed.106.039438. PMID 17475953
- [Background] Dogan H, de Roos A, Geleijins J, Huisman MV, Kroft LJ. The role of computed tomography in the diagnosis of acute and chronic pulmonary embolism. Diagn Interv Radiol. 2015 Jul-Aug;21(4):307-16. doi: 10.5152/dir.2015.14403. PMID 26133321
- [Background] Kim NH, Delcroix M, Jenkins DP, Channick R, Dartevelle P, Jansa P, Lang I, Madani MM, Ogino H, Pengo V, Mayer E. Chronic thromboembolic pulmonary hypertension. J Am Coll Cardiol. 2013 Dec 24;62(25 Suppl):D92-9. doi: 10.1016/j.jacc.2013.10.024. PMID 24355646
- [Background] Lang IM, Pesavento R, Bonderman D, Yuan JX. Risk factors and basic mechanisms of chronic thromboembolic pulmonary hypertension: a current understanding. Eur Respir J. 2013 Feb;41(2):462-8. doi: 10.1183/09031936.00049312. Epub 2012 Jun 14. PMID 22700839
- [Background] Lang IM, Madani M. Update on chronic thromboembolic pulmonary hypertension. Circulation. 2014 Aug 5;130(6):508-18. doi: 10.1161/CIRCULATIONAHA.114.009309. No abstract available. PMID 25092279
- [Background] Lang IM, Simonneau G, Pepke-Zaba JW, Mayer E, Ambroz D, Blanco I, Torbicki A, Mellemkjaer S, Yaici A, Delcroix M. Factors associated with diagnosis and operability of chronic thromboembolic pulmonary hypertension. A case-control study. Thromb Haemost. 2013 Jul;110(1):83-91. doi: 10.1160/TH13-02-0097. Epub 2013 May 16. PMID 23677493
- [Background] van der Bijl N, Klok FA, Huisman MV, van Rooden JK, Mertens BJA, de Roos A, Kroft LJM. Measurement of right and left ventricular function by ECG-synchronized CT scanning in patients with acute pulmonary embolism: usefulness for predicting short-term outcome. Chest. 2011 Oct;140(4):1008-1015. doi: 10.1378/chest.10-3174. Epub 2011 Apr 7. PMID 21474573
- [Background] Klok FA, Zondag W, van Kralingen KW, van Dijk AP, Tamsma JT, Heyning FH, Vliegen HW, Huisman MV. Patient outcomes after acute pulmonary embolism. A pooled survival analysis of different adverse events. Am J Respir Crit Care Med. 2010 Mar 1;181(5):501-6. doi: 10.1164/rccm.200907-1141OC. Epub 2009 Dec 3. PMID 19965808

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CTEPH Patients | Non CTEPH Patients
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CTEPH Patients | Non CTEPH Patients | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (15) | 56 (15) | 58 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 33 | 60
  Male | 23 | 17 | 40
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: To Identify the Accuracy of Routine CTPA for the Distinction of CTEPH From Acute PE.
Description: The sensitivity of CTPA is determined by calculating the proportion of scans that are read as "positive for the CTEPH specific radiological pattern" in patients with confirmed CTEPH and the specificity is determined by calculating the proportion of scans that are read as "negative for the CTEPH specific radiological pattern" in patients without CTEPH.
Time Frame: 1 year
Measure: Mean (95% Confidence Interval); unit: Sensitivity
Arm/Group | CTEPH Patients | Non CTEPH Patients
Number analyzed (Participants) | 50 | 50
Sensitivity | 70 [55 to 82] | 70 [55 to 82]

ADVERSE EVENTS:
Time Frame: 1 year
Description: This was an observational study; no adverse outcomes occured.
Arm/Group | CTEPH Patients | Non CTEPH Patients
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

LIMITATIONS AND CAVEATS:
We studied clear-cut cases of patients with CTEPH and PE patients with RV overload who did not develop CTEPH after 2 years of follow-up, whereas, in clinical practice, the presentation of CTEPH is heterogeneous and the diagnosis is often challenging, for instance, when considering other conditions that may cause PH. Moreover, the prevalence of CTEPH in the cohort was 50%, yet this number is much lower in clinical practice.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-10): https://cdn.clinicaltrials.gov/large-docs/93/NCT03083093/Prot_SAP_000.pdf